CLINICAL TRIAL: NCT01565096
Title: Effect of Adding Vildagliptin on Beta Cell Function and Cardiovascular Risk Markers in Patients With Moderate Metabolic Control During Metformin Monotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ikfe-CRO GmbH (Industry)
Collaborators: Novartis Pharmaceuticals (Industry); IKFE Institute for Clinical Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ikfe-Vilda-001; 2011-004286-32 (EudraCT Number); CLAF237ADE06T (Other: Novartis Pharma GmbH)
Record Dates: First submitted 2012-03-23; First posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Vildagliptin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vildagliptin plus Metformin (Experimental): Metformin (1000 mg BID) + Vildagliptin 50 mg twice daily
  Interventions: Drug: Metformin; Drug: Vildagliptin
- Glimepirid plus Metformin (Active Comparator): Metformin (1000 mg BID) + Glimepiride (individual dosage)
  Interventions: Drug: Metformin; Drug: Glimepiride

INTERVENTIONS:
Drug: Metformin — Metformin 1000 mg BID
  Arms: Vildagliptin plus Metformin
Drug: Metformin — Metformin 1000 mg BID
  Arms: Glimepirid plus Metformin
Drug: Vildagliptin — Vildagliptin 50 mg twice daily
  Arms: Vildagliptin plus Metformin
Drug: Glimepiride — Glimepiride at individual dose
  Arms: Glimepirid plus Metformin

SUMMARY:
The aim of this pilot-study is to investigate the effect of Vildagliptin in comparison to glimepiride on beta cell function and the cardiovascular risk profile in patients previously treated with Metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2
* HbA1c > 6.5%* ≤ 9.5%

  * NOTE: Patients with cardiovascular preconditions (Coronary Heart Disease or Myocard Infarction) require an HbA1c > 7.0% ≤ 9.5%
* Treatment with Metformin at maximal or maximal tolerated dosage, stable for at least 3 months with indication for treatment with an additional medication as judged by the investigator
* Age 30 - 80 years
* Patient consents that his/her family physician will be informed of trial participation

Exclusion Criteria:

* Pre-treatment with insulin, peroxisome proliferator activated receptor (PPAR) gamma agonists or other oral antidiabetic treatments (except Metformin) within the last three months
* History of type-1-diabetes
* Fasting blood glucose >240mg/dl
* Uncontrolled hypertension (systolic blood pressure >160 and/or diastolic blood pressure >90)
* Anamnestic history of acute infections
* Anamnestic history of epilepsy
* Anamnestic history of hypersensitivity to the study drugs or to drugs with similar chemical structures
* History of severe or multiple allergies
* Hereditary galactose intolerance, lapp-lactase defect or glucose-galactose mal-absorption
* Treatment with any other investigational drug within 3 months before trial entry
* Pregnant or lactating women
* Sexually active woman of childbearing age not practicing a highly effective method of birth control as defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal intrauterine devices, sexual abstinence or vasectomized partner
* Progressive fatal disease
* History of drug or alcohol abuse in the past 2 years
* State after kidney transplantation
* Serum potassium > 5.5 mmol/L
* Acute myocardial infarction, open heart surgery or cerebral event (stroke/transient ischemic attack) within the previous 6 months
* Any elective surgery during study participation
* Have had more than one unexplained episode of severe hypoglycemia (defined as requiring assistance of another person due to disabling hypoglycemia) within 6 months prior to screening visit
* History of pancreatitis
* Anamnestic history of dehydration, diabetic precoma or diabetic ketoacidosis
* Acute or scheduled investigation with iodine containing radiopaque material
* Uncontrolled unstable angina pectoris
* Anamnestic history of pericarditis, myocarditis, endocarditis, hemodynamic relevant aortic stenosis, aortic aneurysm or heart insufficiency NYHA III or IV
* Anamnestic recent pulmonary embolism
* History of significant cardiovascular, respiratory, gastrointestinal, hepatic (ALAT and/or ASAT > 3 times the normal reference range), renal (GFR < 60 ml), neurological, psychiatric and/or hematological disease as judged by the investigator
* Lack of compliance or other similar reason that, according to investigator, precludes satisfactory participation in the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Postprandial increase in intact proinsulin levels in patient treated with Vildagliptin and Metformin compared to intact proinsulin levels in patients treated with Glimepiride and Metformin (Area under the curve 0-300 min) | One year

SECONDARY OUTCOMES:
Fasting intact proinsulin levels | One year
Max postprandial intact proinsulin levels | One year
Retinal endothelial response to flicker light stimulation | One year
Mean 24h systolic and diastolic blood pressure | One year
Erythrocyte deformability | One year
E-selectin | One year
Change in body weight | One year
hsCRP | One year
HbA1c | One year
Fasting blood glucose | One year
Number of hypoglycemic events | One year
Adverse events | One year
Drug related adverse events | One year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forst, Prof. Dr., Principal Investigator — Ikfe GmbH
Locations (1):
- ikfe GmbH, Mainz, Germany